CLINICAL TRIAL: NCT03609840
Title: Population Pharmacokinetics and Pharmacodynamics of Thiotepa and TEPA in Pediatric Patients Undergoing Hematopoietic Cell Transplantation (HCT).
Brief Title: Study of Thiotepa and TEPA Drug Exposure in Pediatric Hematopoietic Stem Cell Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 17-21994; 17087 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-01-05; First posted 2018-08-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hematologic Malignancies; Nonmalignant Diseases; Immune Deficiency; Hemoglobinopathies; Genetic Inborn Errors of Metabolism; Fanconi Anemia; Thalassemia; Sickle Cell Disease
Keywords: Thiotepa; TEPA; Pediatric; Hematopoietic; Transplant
MeSH Terms: conditions — Hematologic Neoplasms; Immunologic Deficiency Syndromes; Hemoglobinopathies; Fanconi Anemia; Thalassemia; Anemia, Sickle Cell | interventions — Thiotepa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric Hematopoietic Stem Cell Transplant Recipients: Children undergoing hematopoietic stem cell transplant (HCT) at University of California, San Francisco Benioff Children's Hospital
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — Given IV
  Other Names: Alkylating antineoplastic agent; Tepadina

SUMMARY:
Thiotepa is a chemotherapy drug used extensively in bone marrow transplantation. Thiotepa is a prodrug that undergoes metabolic conversion in the liver by CYP2B6 and CYP3A4 to its primary active metabolite, triethylene phosphoramide (TEPA). The goal of this study is to determine what causes some children to have different drug concentrations of thiotepa and TEPA in their bodies and if drug levels are related to whether or not a child experiences severe side-effects during their bone marrow transplant. The hypothesis is that certain clinical and genetic factors cause changes in thiotepa and TEPA drug levels in pediatric bone marrow transplant patients and that high levels may cause severe side-effects.

DETAILED DESCRIPTION:
Thiotepa is an alkylating agent with potent antitumor and immunosuppressive properties used in conditioning regimens of pediatric hematopoietic cell transplantation (HCT) to promote stem cell engraftment. Thiotepa is a prodrug that undergoes metabolic conversion in the liver by CYP2B6 and CYP3A4 to its primary active metabolite, TEPA.

This is a single-center, prospective, non-interventional pharmacokinetics (PK) study investigating the clinical pharmacology of thiotepa and TEPA in 60 children undergoing hematopoietic stem cell transplant (HCT) at University of California, San Francisco Benioff Children's Hospital. Patients would receive thiotepa regardless of whether or not they decide to consent to PK sampling.

Thiotepa doses will not be adjusted based on PK data. The investigators will apply the combination of a limited sampling strategy and population PK methodologies to determine specific factors influencing thiotepa and TEPA exposure in pediatric HCT recipients. Population PK methodologies support the use of sparse sampling and therefore allow the investigators to investigate drug levels in a pediatric population that would otherwise not be feasible using traditional intensive PK sampling.

Subjects will undergo PK sampling of plasma thiotepa and TEPA drug concentrations over the duration of thiotepa therapy (3 to 5 days).

To evaluate sources of variability impacting thiotepa and TEPA exposure clinical data will be obtained from the patient's medical chart on each day of PK sampling.

A single blood draw for the collection of DNA and genotyping of single nucleotide polymorphisms of genes involved in fludarabine activation, transport or elimination will occur in all patients.

To assess exposure-response relationships neutrophil engraftment, treatment-related toxicity, and survival data will be collected through day 100 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. be between 0 to 17 years of age;
2. meet protocol specific eligibility criteria for autologous or allogeneic HCT
3. will be receiving thiotepa as part of their conditioning regimen.

Exclusion Criteria:

* Any child 7-17 years of age unwilling to provide assent
* Parent or guardian unwilling to provide written consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population for the proposed study includes children 0-17 years of age undergoing autologous and allogeneic HCT for the treatment of malignant and nonmalignant disorders. Patients receiving thiotepa over 3 to 5 days are eligible to participate. All patients enrolled in this study will undergo PK sampling on the inpatient pediatric BMT unit at UCSF Benioff Children's Hospital. The proposed research will not study any patients receiving thiotepa in a clinic or any other out-patient setting.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of thiotepa for HCT in pediatric patients. | 2 hours post start of infusion
  Area-under-the-curve (AUC) will be derived from the empirical Bayes estimates of individual clearance
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of thiotepa for HCT in pediatric patients. | 4 hours post start of infusion
  Area-under-the-curve (AUC) will be derived from the empirical Bayes estimates of individual clearance
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of thiotepa for HCT in pediatric patients. | 6 hours post start of infusion
  Area-under-the-curve (AUC) will be derived from the empirical Bayes estimates of individual clearance
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of thiotepa for HCT in pediatric patients. | 24 hours post start of infusion
  Area-under-the-curve (AUC) will be derived from the empirical Bayes estimates of individual clearance

SECONDARY OUTCOMES:
Event free survival according to the AUC of thiotepa | 1 month post transplant
  Death due to any cause within 1 month post-transplant will be considered an event.
Event free survival according to the AUC of thiotepa | 3 months post transplant
  Death due to any cause within day 3 months post-transplant will be considered an event.
Event free survival according to the AUC of thiotepa | 1 year post transplant
  Death due to any cause within day 1 year post-transplant will be considered an event.

CONTACTS AND LOCATIONS:
Overall Officials: Janel Long-Boyle, PharmD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No